CLINICAL TRIAL: NCT07340554
Title: Neuroimaging of Instrumental Learning Networks in Adolescent Cannabis Use Treatment
Brief Title: Neuroimaging of Adolescent Cannabis Use Treatment
Acronym: ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joseph Aloi, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27183; K23DA063832 (NIH)
Record Dates: First submitted 2026-01-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use; Cannabis Dependence; Cannabis Use Disorder; Cannabis Abuse; Cannabis Intoxication; Cannabis Smoking; Cannabis Withdrawal; Cannabis-Related Disorder; Cannabis Abuse, in Remission; Cannabis Abuse, Episodic Use; Marijuana; Marijuana Abuse; Marijuana Use; Marijuana Smoking; Marijuana Dependence; Marijuana User; Marijuana-Related Disorder; Marijuana Use Disorder; Addiction; Addiction, Substance; Substance Use; Substance Use Disorders; Substance Dependence; Substance Abuse; Substance Related Problem; Substance Abuse Drug Chronic
Keywords: Cannabis; Marijuana; Addiction
MeSH Terms: conditions — Marijuana Abuse; Marijuana Smoking; Marijuana Use; Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Contingency Management and Elastic Net Regression (Other): All participants will receive Contingency Management treatment for Cannabis Use.
  An elastic net regression model will be applied to the neuroimaging data for all participants to estimate scores on the CUDIT.
  Interventions: Behavioral: Contingency Management; Device: Elastic Net Regression

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management is an evidence-based behavioral intervention used to treat substance use disorders, including cannabis use disorder (CUD). Contingency management operates on the principles of instrumental learning, where positive reinforcement is used to encourage desired behaviors, such as abstinence from cannabis. First, specific target behaviors are identified for reinforcement. In CUD, this is often abstinence from cannabis use, verified through regular urine drug screens and self-reports. If the target behavior (i.e., abstaining from cannabis for a specified time period) is achieved, then patients receive tangible rewards immediately after attaining the target behavior. These rewards are often in the form of money, vouchers, or other incentives that are meaningful to the individual. We will examine whether success during contingency management treatment for cannabis use is associated with neural activity during instrumental learning in N=80 adolescents ages 14-17.
Device: Elastic Net Regression — We will apply an elastic net regression model to the neuroimaging data to estimate CUDIT score based on neuroimaging data.

SUMMARY:
This study is testing whether brain activity related to learning can help predict how well teens respond to a treatment program designed to reduce cannabis use. Teens ages 14-17 will complete a brain scan and then take part in 10 weekly virtual sessions where they report cannabis use and complete drug tests at home. Participants can earn prizes for staying cannabis-free.

DETAILED DESCRIPTION:
This is a 13-week clinical trial to examine whether success during contingency management treatment for cannabis use is associated with baseline functioning of instrumental learning neuro-circuitries. The investigators propose to recruit N=80 youths ages 14-17 with varying levels of cannabis use. Following phone prescreening, participants will undergo informed consent/assent and eligibility assessment with an in-person visit. Participants who are eligible will undergo a functional magnetic resonance imaging (fMRI) scan where participants will perform an instrumental learning task during a second in-person visit. At this visit, participants and participants' guardians or most recent caregiver will be provided with ten urine drug screens. A tutorial will be provided by study staff on how to administer and read urine drug screens. After the fMRI scan, participants will undergo ten weekly virtual contingency management sessions administered via HIPAA-compliant telehealth software (e.g., Microsoft Teams). At each contingency management session, participants will be asked to provide a urine sample, and participants' guardians will be asked to administer the urine drug screen based on this sample. At each contingency management session, the timeline followback will be used to assess which days since the last session participants used cannabis at all. Finally, at each contingency management session, participants will answer brief questionnaires regarding participants' current cannabis cravings and cannabis withdrawal symptoms. For the first two sessions, participants will be able to spin a virtual wheel to win prizes (either positive affirmations or amazon gift cards in varying amounts from $5-$100) for producing a urine drug screen and answering the questions. For sessions 3-10, participants will spin the virtual wheel to win prizes after producing a urine drug screen that is negative for cannabinoids and reporting that they have not used cannabis since the last session. After the ten weekly contingency management sessions, participants will return for an in-person visit where participants will answer questions regarding their cannabis use disorder symptoms during the contingency management treatment and readiness to change. The investigators' specific aims are to identify associations between baseline Cannabis Use Disorder (CUD) symptom levels and neural activity during instrumental learning in cannabis-using adolescents (Aim 1) and Identify associations between neural activity during instrumental learning and reductions in cannabis use frequency during contingency management (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* 14-17 year old youth
* Guardian 18 years or older
* Youth is MRI-eligible: No metal implants, prosthetics, orthodontic devices, transdermal medication patches, piercings and/or hair or eyelash extensions that cannot easily be removed, metallic ink tattoos on the neck or face, or claustrophobia, and are not pregnant
* Youth must endorse having used cannabis at least once per week over the past month

Exclusion Criteria:

* Youth has a history of Fetal Alcohol Spectrum Disorder, intellectual disorders, pervasive development disorder or autism spectrum disorder, psychotic disorders, history of neurological problems (epilepsy, traumatic brain injury, brain tumor, cerebrovascular disease) by parent/guardian report
* Youth or caretaker who is monolingual non-English speaker
* Youth who is currently experiencing active psychosis symptoms or suicidal/homicidal ideation or who has been hospitalized within the past 6 months for psychosis or suicidality/homicidality
* Youth who is currently undergoing contingency management treatment for cannabis use disorder

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Cannabis use frequency | Past 30 days
  The investigators will measure cannabis use frequency via percent of days where cannabis was used over the past 30 days via the Timeline Followback Scale (Sobell and Sobell, 1992)
Cannabis Use Disorder Identification Test (CUDIT) Score | Baseline
  The CUDIT (Adamson et al., 2010) is a measure of cannabis use disorder symptom level. This scale is an 8-item scale that asks about cannabis use disorder symptoms over the past year and is scored on a scale of 0 (no cannabis use in the past year) to 32 (daily cannabis use, physical and psychological dependence symptoms, severe cannabis misuse). The CUDIT will be measured once at the baseline screening visit.

SECONDARY OUTCOMES:
Total quantity of cannabis use | Past 30 days
  The investigators will measure cannabis use quantity via the Timeline Followback Scale (Sobell and Sobell, 1992). For each day participants report cannabis use on the Timeline Followback Scale, participants will be asked to estimate the number of grams of cannabis used.
Cannabis withdrawal | 12 weeks
  Cannabis withdrawal will be measured at 12 different time points via the Cannabis Withdrawal Scale (Milin, Manion, Dare, and Walker, 2008). The Cannabis Withdrawal Scale is a 16-item scale that evaluates cannabis withdrawal symptoms, such as sleep difficulties, nervousness, anxiety, tension, and cravings for cannabis. This scale will be administered at the scanning visit, each of the 10 contingency management visits, and at the follow-up visit.
Cannabis expectancy | 12 weeks
  Cannabis expectancy will be measured at 2 time points via the Marijuana Effects Expectancy Scale-Brief (Torrealday et al., 2008). The Marijuana Effects Expectancy Scale-Brief is a six item scale that measures expected effects (relaxation, reduced anxiety, cravings) of marijuana use. This scale will be administered at the scanning visit and the follow-up visit.
Proportion of negative cannabis urine drug screen | 12 weeks
  Urine drug screens will be collected at each visit (13 total). The investigators will track the proportion of urine drug screens that are negative over all visits and that are negative over the 10 contingency management visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States